CLINICAL TRIAL: NCT01908907
Title: Bridging the Docosahexaenoic Acid (DHA) Gap: The Effects of Omega-3 Fatty Acid Supplementation in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHA Gap
Record Dates: First submitted 2013-07-02; First posted 2013-07-26 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Prematurity
Keywords: Premature Infants; DHA(docosahexaenoic acid); DHA deficit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA oil (Active Comparator): DHA oil administered 50 mg/d (0.18ml)as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  Interventions: Dietary Supplement: DHA oil
- (MCT) control oil (Placebo Comparator): MCT oil administered 0.18ml as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  Interventions: Dietary Supplement: (MCT) Control oil

INTERVENTIONS:
Dietary Supplement: DHA oil — Therapy Group:DHA oil administered at 50 mg/d (0.18ml) as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  Arms: DHA oil
Dietary Supplement: (MCT) Control oil — Placebo Group:MCT oil administered at 0.18 ml as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  Arms: (MCT) control oil

SUMMARY:
The purpose of this study is to understand if the "DHA gap" can be corrected by giving a daily dose of DHA oil to preterm babies.

DHA is an essential omega-3 fatty acid, which means our body cannot make DHA. We have to take it in through our diet. DHA is important for normal brain and eye health and it may also decrease inflammation. This is important for premature babies because they are at a greater risk for getting diseases related to inflammation, especially in their lungs, eyes and intestines. Since DHA is so important for normal growth, you will find DHA naturally in breast milk and it is now added to infant formula. But the amount in breast milk and infant formula is about half of what your infant should expect to get in the womb (about 13-29mg per day in breast milk vs. 50-75mg per day in the womb). Very premature babies are at an even greater disadvantage because they cannot always eat very much right away and that is the only way they can get essential fatty acids in their body. This means premature babies are getting less DHA than they would in the womb and then the "DHA gap" continues for a longer period of time. This gap also comes at a time when their brain is growing most rapidly and their bodies need it the most. This trial is designed to see if giving DHA, even before the baby can take food orally, will raise his/her DHA blood levels to those of normal term babies.

DETAILED DESCRIPTION:
Docosahexaenoic acid (DHA) is an essential fatty acid (FA) important for health and neurodevelopment. Premature infants are at risk of DHA deficiency and circulating levels directly correlate with health outcomes. Most supplementation strategies have focused on increasing DHA content in mother's milk or infant formula. However, extremely premature infants may not reach full feedings for weeks and commercially available parenteral lipid emulsions do not contain preformed DHA, so blood levels decline rapidly after birth. Our objective is to develop a DHA supplementation strategy to overcome these barriers. This single-center, double-blind, randomized, controlled trial determined feasibility, tolerability and efficacy of daily enteral DHA supplementation (50 mg/day) in addition to standard nutrition for preterm infants (24-34 weeks gestational age) beginning in the first week of life. Blood FA levels will be analyzed at baseline, full feedings and near discharge in DHA or placebo supplemented preterm infants. Term peers will also have blood FA levels analyzed for comparison. Growth, feeding tolerance and adverse outcomes (NEC, intraventricular hemorrhage (IVH), thrombocytopenia, sepsis) will be evaluated. Study progress and safety will be monitored by an external Data Safety Monitoring Board (DSMB). Overall, the study aims to determine if daily enteral DHA supplementation is feasible and alleviates deficiency in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 24 and 33 6/7 weeks gestation
* must be less than or equal to 1 week of age

Exclusion Criteria:

* infants who are considered by the medical team to be non-viable
* infants with multiple or severe congenital anomalies such as gastroschisis, congenital chylothorax or other illnesses that do not allow a feeding tube to be placed or utilized at 7 days of age.
* term infants: who are born to mothers with diabetes or are small for gestational age (SGA-less than the 10th% for adjusted gestational age
* All families consented for this study will need to be able to read and write English
* Mother must be 18 years of age or older
* Taking Omegaven

Ages: 24 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Baack, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Health USD, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. All data is de-identified for review by DSMB or others.

REFERENCES:
- [Derived] Baack ML, Puumala SE, Messier SE, Pritchett DK, Harris WS. Daily Enteral DHA Supplementation Alleviates Deficiency in Premature Infants. Lipids. 2016 Apr;51(4):423-33. doi: 10.1007/s11745-016-4130-4. Epub 2016 Feb 4. PMID 26846324
- [Derived] Baack ML, Puumala SE, Messier SE, Pritchett DK, Harris WS. What is the relationship between gestational age and docosahexaenoic acid (DHA) and arachidonic acid (ARA) levels? Prostaglandins Leukot Essent Fatty Acids. 2015 Sep;100:5-11. doi: 10.1016/j.plefa.2015.05.003. Epub 2015 Jun 17. PMID 26205427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety infants, less than or equal to one week of age, were recruited from the Sanford Health Boekelheide Neonatal Intensive Care Unit (NICU) between October 2012 and March 2014.
Pre-assignment Details: Preterm infants were between 24 and 33 6/7 weeks gestational age (GA) at birth. Adaptive enrollment was used to assure that infants <28 weeks GA were enrolled over the same time period as more commonly admitted preterm infants >28 weeks GA.
Groups:
- DHA Oil: DHA oil administered 50 mg/d (0.18ml)as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  DHA oil administered at 50 mg/d (0.18ml) Or MCT oil administered at 0.18 ml
- Medium Chain Triglyceride (MCT) Control Oil: MCT oil administered 0.18ml as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  Placebo Group:MCT oil administered at 0.18 ml as an oil emulsion
Period: Overall Study
Arm/Group | DHA Oil | Medium Chain Triglyceride (MCT) Control Oil
Started | 31 | 29
Completed | 29 | 29
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Preterm infants less than one week of age and born between 24 and 33 6/7 week GA were randomized to receive 50mg/d of enteral DHA
Groups:
- DHA Supplemented: Preterm infants (31) randomized to receive 50mg/d of enteral DHA supplementation
- Placebo Supplemented: Preterm infants (29) randomized to receive placebo study oil
- Total: Total of all reporting groups
Arm/Group | DHA Supplemented | Placebo Supplemented | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: weeks of GA] | 30.69 (2.42) | 30.35 (2.46) | 30.52 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 16 | 14 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 0 | 0
  Non-Hispanic | 28 | 25 | 53
  Unknown | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Days to Reach Full Enteral Feedings and Days on Study Oil.
Description: This study was designed to determine feasibility and tolerability of enteral DHA supplementation, but was not intended to determine the effects of DHA on health related outcomes. Tolerability was measured by days to reach full enteral feedings, days on study oil, GA at completion of the study and postnatal growth. The days to reach full enteral feedings was defined as enteral intake of 100kcal/kg/d. Safety and tolerability was closely monitored under the oversight of an independent DSMB.
Time Frame: From enrollment until the infant reaches full feed or is discharged from the NICU, whichever comes first, assessed up to 50 days.
Population: Comparison between preterm groups that received either DHA oil or MCT (placebo control) oil were made.
Measure: Mean (Standard Deviation); unit: days
Groups:
- (MCT) Control Oil: MCT oil administered 0.18ml as an oil emulsion enterally with feedings or by gavage tube if the infant has one.
  Placebo Group:MCT oil administered at 0.18 ml as an oil emulsion
Arm/Group | DHA Oil | (MCT) Control Oil
Number analyzed (Participants) | 31 | 29
days
  Days to reach full enteral feedings | 20.00 (8.32) | 16.21 (7.41)
  Days on Study oil | 34.00 (19.2) | 33.71 (16.32)
Statistical Analysis 1: Comparison: DHA Oil vs (MCT) Control Oil; All analyses used the intent-to-treat study population. A linear mixed model was used to assess differences in time to full feeds, days on study drug, and gestational age at discharge. These models included a random effect for multiples, which was maintained in the model after testing. Fixed effects included treatment and GA group for time to full feeds and days on study drug and treatment effect for gestational age at discharge; Test type: Superiority or Other; p = 0.07, Regression, Linear; Outcome was transformed using a natural logarithm transformation. Models included gestational age group since the randomization was blocked; Median Difference (Net) = 13.5, 95% CI 2-sided [0.2 to 28.7], Standard Error of Mean 6.5 — Since analyzed on the log scale, estimates provide are % change rather than absolute change between group

2. Primary Outcome: Feasibility and Tolerability of Daily Enteral DHA Oil - Weight Change
Description: A linear mixed model was used to explore weight over time.
Time Frame: 30 days from birth
Population: Comparison between preterm groups that received either DHA oil or MCT (placebo control) oil were made. They had DHA levels measured to be used as a reference population in our NICU.
Measure: Mean (Standard Error); unit: Grams per day
Groups:
- DHA Supplemented: Preterm infants supplemented with 50mg/d (0.18ml) of enteral DHA from the first week of life until term GA or discharge, whichever came first.
- MCT (Placebo Control Group): Preterm infants receiving 0.18 ml of MCT (control oil) from the first week of life until term GA or discharge, whichever came first.
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
Grams per day | 18.4 (0.57) | 18.4 (0.57)
Statistical Analysis 1: Comparison: DHA Supplemented vs MCT (Placebo Control Group); Linear mixed models were used to explore growth over time (weight, length and head circumference). These models included a random effect for intercepts and slopes to account for subject specific growth over time as well as a random effect for possible correlation between twins and triplets present in the data set. Fixed effects included both a linear and quadratic time effect, GA at birth, treatment group, full feeds (yes/no), and interactions. Non-significant interactions were eliminated; Test type: Superiority or Other; p = 0.048, Regression, Linear; This is a complex regression model including linear and quadratic growth and interactions as specified above; Mean Difference (Net) = 0.016, Standard Error of Mean 0.008

3. Primary Outcome: Long Chain Polyunsaturated Fatty Acid (LCPUFA) Levels - Docosahexaenoic Acid (DHA) Levels in Whole Blood
Description: Linear mixed models were also used to examine the association between each FA of interest and treatment group over time. Since only three time points were available for FA measurement, only a random intercept was included in the models. For these models, the random effect for multiples was again found to be not needed and removed. Primary outcome variables for this analysis included LNA, ALA, ARA and DHA. Only early/late preterm status was included in the model as a covariate since this was a stratification variable. Continuous dependent variables were transformed using the natural logarithm as needed to meet the assumptions of the regression model (this included LNA and ALA).
Time Frame: At baseline (enrollment, < 1 week of age), full feedings, discharge
Measure: Mean (Standard Deviation); unit: mol% (composition) of fat
Groups:
- DHA Supplemented: Preterm infants supplemented with 50mg/d (0.18ml) of enteral DHA from the first week of life until term GA or discharge, whichever came first.
  LCPUFA levels were measured at baseline, after reaching full enteral feedings and at discharge or term GA, whichever came first.
- MCT (Placebo Control Group): Preterm infants receiving 0.18 ml of MCT (control oil) from the first week of life until term GA or discharge, whichever came first.
  LCPUFA levels were measured at baseline, after reaching full enteral feedings and at discharge or term GA, whichever came first.
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
mol% (composition) of fat
  Baseline Comparisons | 2.91 (0.45) | 2.88 (0.68)
  Full Enteral Feedings | 2.83 (0.50) | 3.03 (0.54)
  Discharge | 2.87 (0.50) | 3.55 (0.44)

4. Primary Outcome: Feasibility and Tolerability of Daily Enteral DHA Oil - Length Change
Description: A linear mixed model was used to explore length over time.
Time Frame: 30 days from birth
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Centimeters per day
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
Centimeters per day | 0.13 (0.006) | 0.12 (0.004)

5. Primary Outcome: Feasibility and Tolerability of Daily Enteral DHA Oil - Head Circumference
Description: A linear mixed model was used to explore head circumference over time.
Time Frame: 30 days from birth
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Centimeters per day
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
Centimeters per day | 0.10 (0.004) | 0.10 (0.004)

6. Secondary Outcome: LCPUFA Levels - Arachidonic Acid (ARA) in Whole Blood
Description: as for outcome 3
Time Frame: At baseline (enrollment, <1 week of age), full feedings and discharge
Measure: Mean (Standard Deviation); unit: wt:wt% of total fat in sample
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
wt:wt% of total fat in sample
  Baseline | 13.21 (2.22) | 14.89 (1.89)
  Full Enteral Feedings | 14.35 (1.51) | 14.87 (1.50)
  Discharge | 14.31 (1.26) | 13.94 (1.67)

7. Other Pre Specified Outcome: LCPUFA Levels - Alpha-linolenic Acid (ALA) in Whole Blood
Description: as for outcome 3
Time Frame: Baseline (<1 week of age), full enteral feedings and discharge
Measure: Mean (Standard Deviation); unit: wt:wt% (composition) of total fat
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
wt:wt% (composition) of total fat
  Baseline | 0.74 (0.50) | 0.55 (0.33)
  Full enteral feedings | 0.21 (0.13) | 0.20 (0.11)
  Discharge | 0.24 (0.13) | 0.26 (0.13)

8. Other Pre Specified Outcome: LCPUFA Levels - Linoleic Acid (LNA)
Description: as for outcome 3
Time Frame: Baseline, full feedings and discharge
Measure: Mean (Standard Deviation); unit: wt:wt% (composition) of fat in sample
Arm/Group | DHA Supplemented | MCT (Placebo Control Group)
Number analyzed (Participants) | 31 | 29
wt:wt% (composition) of fat in sample
  Baseline | 18.45 (4.51) | 16.45 (3.39)
  Full feedings | 14.72 (2.05) | 14.95 (2.04)
  Discharge | 15.37 (2.39) | 16.64 (3.18)

ADVERSE EVENTS:
Time Frame: Monitored for 30 days after last dose of study medication.
Arm/Group | DHA Oil | (MCT) Control Oil
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/29
Other Adverse Events (participants affected / at risk) | 31/31 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DHA Oil (N=31) | (MCT) Control Oil (N=29)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DHA Oil (N=31) | (MCT) Control Oil (N=29)
Bronchopulmonary Dysplasia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sepsis (Grade 4) (Infections and infestations) | 3 (3) | 3 (3)
Retinopathy of Prematurity (Eye disorders) | 7 (7) | 5 (5)
Gastro-esophageal Reflux Disease (Gastrointestinal disorders) | 6 (6) | 4 (4)
Milk Soy Protein Intolerance (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Intraventricular Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Periventricular Leukomalacia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 20 (20) | 14 (14)
Apnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Other Blood and lymphatic disorders (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Other Cardiac Disorders (Cardiac disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (2)
Congenital heart defect (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysfunctional bottling/swallowing (Gastrointestinal disorders) | 7 (7) | 1 (1)
Other Endocrine Disorders (Endocrine disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorder NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other General Disorder (General disorders) | 2 (2) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other Infections and Infestations (Infections and infestations) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Other Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Other Musculoskeletal Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Patent Ductus Arteriosus (Cardiac disorders) | 3 (3) | 3 (3)
Periodic Breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Physiologic murmur (Cardiac disorders) | 13 (15) | 6 (7)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Other Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other Skin Disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Other Vascular Disorders (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No